CLINICAL TRIAL: NCT07308574
Title: Multicenter, Open-label, Single-arm, Post-Marketing Clinical Study to Evaluate the Efficacy and Safety of Ravulizumab in Participants Clinically Diagnosed as Atypical Hemolytic Uremic Syndrome
Brief Title: Post-Marketing Clinical Study of Ravulizumab in Participants With Clinical aHUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D928BL00001; NEPH-ULT-501 (Registry Identifier: Alexion)
Record Dates: First submitted 2025-12-17; First posted 2025-12-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: aHUS; Atypical Hemolytic Uremic Syndrome
Keywords: aHUS; atypical hemolytic uremic syndrome; ravulizumab
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): Participants will receive a weight-based loading dose of ravulizumab, followed by a weight-based dose 2 weeks after loading dose administration, then weight-based maintenance doses every 8 weeks via intravenous (IV) infusion.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive ravulizumab via IV infusion.

SUMMARY:
The primary objective of this study is to assess the platelet count response to ravulizumab in participants clinically diagnosed as atypical hemolytic uremic syndrome (aHUS).

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥20 kilograms (kg)
* Participants clinically diagnosed as aHUS who have any of diseases/conditions listed below (including participants in whom Thrombotic microangiopathy (TMA) has not been improved even after treatment for the pathogenesis of diagnosed secondary TMA and therefore, diagnosis of aHUS was made).
* Infection (except for pneumococcal infection and Siga toxin-producing Escherichia coli infection)
* During pregnancy or postpartum
* Post-renal transplantation
* Hypertensive crisis/malignant hypertension
* Systemic lupus erythematosus and related diseases (e.g. dermatomyositis, mixed connective tissue disease, etc.)
* Participants with the following three signs:
* Thrombocytopenia: Platelet count <150,000/microliter (μL)
* Microangiopathic haemolytic anaemia: Hb < 10 grams per deciliter (g/dL) (*)
* Acute kidney injury: one of the following is fulfilled; 1. ΔsCr ≥ 0.3 milligrams per deciliter (mg/dL) (within 48 hours), 2. 1.5-fold increase from baseline sCr (within 7 days), 3. urinary output ≤ 0.5 mL/kg/hour for ≥ 6 hours.
* No prior treatment with complement inhibitors.
* The investigator plans to provide the participant with 26-week treatment with ravulizumab in accordance with the treatment policy in clinical practice.
* Ravulizumab treatment is planned to be initiated within 14 days after onset of the latest TMA episode.
* Participants consenting to meningococcal vaccine administration and appropriate antibiotic prophylaxis (if required).

Exclusion Criteria:

* Participants with TTP, STEC-HUS, secondary TMA that is obviously unrelated to complement abnormality.
* Participants with TMA caused by malignant tumors, abnormal Cobalamin C metabolism, Streptococcus pneumoniae, drugs, autoimmune diseases other than systemic lupus erythematosus and related diseases (e.g. scleroderma etc.), or hematopoietic stem cell transplantation
* Participants with pathological complement gene variants (CFH, CFI , CD46 (MCP), C3, CFB, THBD, DGKE) associated with the development of aHUS at enrolment
* Participants with positive anti-factor H antibodies
* More than 14 day from onset of TMA to the planned start of ravulizumab treatment
* Chronic kidney disease or irreversible renal impairment that requires chronic dialysis
* Presence of unresolved meningococcal disease
* Judgement by the investigator that the participant is not eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Showing Improvement in Platelet Count During the 26-week Ravulizumab Treatment | Baseline up to Week 26

SECONDARY OUTCOMES:
Percentage of Participants Showing Improvement in Renal Function During the 26-week Ravulizumab Treatment | Baseline up to Week 26
Percentage of Participants Showing Improvement in Platelet Count | Day 4 and on Weeks 1, 2, 10, 18, and 26
Percentage of Participants Showing Improvement in Renal Function | Day 4 and on Weeks 1, 2, 10, 18, and 26
Percentage of Participants Showing Improvement in Complete Thrombotic Microangiopathy (TMA) Response or Partial TMA Response | Day 4 and on Weeks 1, 2, 10, 18, and 26
Percentage of Participants who are on Dialysis on Day 1 and are Able to Withdraw From Dialysis by Week 26 | Baseline (Day 1) up to Week 26
Change from Baseline in Platelet Count | Baseline (Day 1), Week 26
Change From Baseline in Hemoglobin | Baseline (Day 1), Week 26
Change From Baseline in Lactate Dehydrogenase | Baseline (Day 1), Week 26
Change From Baseline in Estimated Glomerular Filtration Rate | Baseline (Day 1), Week 26

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (12):
  - Research Site, Bunkyō City
  - Research Site, Hirakata-shi
  - Research Site, Iruma-Gun
  - Research Site, Kyoto
  - Research Site, Matsumoto-shi
  - Research Site, Miyazaki
  - Research Site, Nagoya
  - Research Site, Nara
  - Research Site, Nerima-ku
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Tsu

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR